CLINICAL TRIAL: NCT04630184
Title: Development and Impact of a Virtual Reality Exposure Intervention on Social Physical Anxiety During Physical Activity in Women With Obesity
Brief Title: A Virtual Reality Exposure Intervention on Social Physical Anxiety in Women With Obesity
Acronym: SPA-VR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universite du Quebec en Outaouais (Other)
Responsible Party: Principal Investigator, Aurelie Baillot, Professor, Universite du Quebec en Outaouais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Record Dates: First submitted 2020-11-03; First posted 2020-11-16 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Obesity; Exercise; Virtual Reality
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The reserarch assistant (for assesement) will be blind of the group allocation, as well as the kinesiologist (but not the psychologist).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality and exercice (Experimental): This group will receive the exposure intervention in virtual reality and physical activity during 12 weeks
  Interventions: Behavioral: Exposure intervention in virtual reality; Behavioral: Exercise
- Placebo and exercice (Placebo Comparator): This group will receive the placebo intervention (relaxation) and physical activity during 12 weeks
  Interventions: Behavioral: Exercise; Behavioral: Placebo
- waiting list (No Intervention): This group will receive no intervention during 12 weeks, then will be randomized in the experimental or placebo group

INTERVENTIONS:
Behavioral: Exposure intervention in virtual reality — 6 sessions of 45 minutes weekly and 2 follow-up meetings (3 and 6 weeks after the weekly follow-up) with cognitive restructuring and VR exposure supervised by psychologists
  Arms: Virtual reality and exercice
Behavioral: Exercise — Participants will have to go twice a week, for 12 weeks to carry out 2 individual endurance training sessions of 45 minutes (moderate to vigorous intensity), supervised by a kinesiologist. Participants will also have to complete a 3rd 60-minute endurance session at home (or two 30-minute sessions).
  Arms: Placebo and exercice; Virtual reality and exercice
Behavioral: Placebo — 6 sessions of 45 minutes weekly and 2 follow-up meetings (3 and 6 weeks after the weekly follow-up) Discussion around social physical anxiety, stress management (relaxation and breathing) supervised by psychologists
  Arms: Placebo and exercice

SUMMARY:
The objectives of the project are to: i) assess the feasibility and acceptability of the protocol and the VR exposure intervention in women with obesity, and ii) obtain an estimate of the effect of VR exposure intervention associated with an exercise training on SPA, compliance, adherence and persistence to the exercise training, as well as persistence in PA practice in the middle term to calculate the sample size for a future larger randomized controlled trial (RCT) in women with obesity.

A RCT of feasibility will be carried out. Forty-five women with obesity and a high level of SPA will be randomized into one of the following three groups: 1) Exercice and VR exposure (Ex + expo), 2) Exercise and psychological intervention control (Ex + control) or 3) waiting list (WL).

The interventions will have a physical exercise training (identical for all) and a psychology intervention (different according to the condition: VR exposure or control). The feasibility and acceptability of the protocol and the VR exposure intervention will be assessed at the end of the study. SPA, PA practice, anthropometry, internalization of weight bias, body appreciation, perceived pleasure, motivational regulation, self-efficacy, affects as well as perception effort will be evaluated with questionnaires and scales validated before and after the intervention and 6 months after the end of the intervention. Sociodemographic data, depressive symptoms, problematic eating behaviors and propensity to immersion will be assessed during the initial visit only. Adherence, adherence and persistence to the PA program will be calculated at the end of the intervention. Persistence in PA practice will be calculated using data collected immediately after the end of the intervention and 6 months after the intervention.

DETAILED DESCRIPTION:
Several studies show that a high level of social physical anxiety (SPA) can lead to avoidance and poor adherence to physical activity (PA) programs. Although this link is known and a high level of SPA is frequently found in women with obesity, no psychological intervention specific to the treatment of SPA has been developed to date. Exposure therapy is the treatment of choice for general social anxiety. However, this format of therapy can cause great discomfort for the patient and prevents complete control of the environment by the clinician. Virtual reality (VR), commonly employed in the treatment of anxiety disorders, offers a solution to these problems by allowing exposure to human stimuli in an adaptable environment and under the control of the clinician, with a reduction in stress patient discomfort.

The objectives of the project are to: i) assess the feasibility and acceptability of the protocol and the VR exposure intervention in women with obesity, and ii) obtain an estimate of the effect of VR exposure intervention associated with an exercise training on SPA, compliance, adherence and persistence to the exercise training, as well as persistence in PA practice in the middle term to calculate the sample size for a future larger randomized controlled trial (RCT) in women with obesity.

A RCT of feasibility will be carried out. Forty-five women with obesity and a high level of SPA will be randomized into one of the following three groups: 1) Exercice and VR exposure (Ex + expo), 2) Exercise and psychological intervention control (Ex + control) or 3) waiting list (WL).

The interventions will have a physical exercise training (identical for all) and a psychology intervention (different according to the condition: VR exposure or control). The feasibility and acceptability of the protocol and the VR exposure intervention will be assessed at the end of the study. SPA, PA practice, anthropometry, internalization of weight bias, body appreciation, perceived pleasure, motivational regulation, self-efficacy, affects as well as perception effort will be evaluated with questionnaires and scales validated before and after the intervention and 6 months after the end of the intervention. Sociodemographic data, depressive symptoms, problematic eating behaviors and propensity to immersion will be assessed during the initial visit only. Adherence, adherence and persistence to the PA program will be calculated at the end of the intervention. Persistence in PA practice will be calculated using data collected immediately after the end of the intervention and 6 months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* woman
* inactive (<150 min. of moderate to vigorous PA / week )
* aged between 18 and 45 years
* BMI ≥ 30 kg / m2
* to be able to go to Université du Québec en Outaouais twice a week

Exclusion Criteria:

* to have a low to moderate social physical anxiety level (SPA score <27/45 on the physical and social anxiety scale )
* suffer from hypersensitivity to motion sickness
* to be pregnant or plan to become over the next year
* to take medication that may influence weight
* to have undergone bariatric surgery
* to have a contraindication to physical activity
* to have participated in a physical activity program in the last 6 months supervised
* to have an intellectual disability, and have a severe and persistent psychiatric problem (psychosis, bipolar disorder).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the protocol and the intervention | At the end of the study (+ 36 weeks)
  The feasibility of the protocol will be assessed at the end of the study using the following criteria: i) the recruitment rate (number of participants recruited per month), ii) the retention rate (number of participants who have completed all the assessments and focus group and reason for dropout), iii) percentage of missing data (number of missing data out of number of total data) and iv) acceptance of randomization.
  The feasibility of the intervention will be evaluated at the end of the study using the following criteria: v) the participation rate (number of eligible participants who agreed to participate in the study), vi) the participation rate adherence (number of participants who completed the 8 psychological intervention sessions), vii) the attrition rate (number of participants who abandoned the psychological intervention and reasons).
  The achievement of the following criteria will be considered as a success factor in terms of feasibility (14, 23): i) recruitment rate ≤ 5.6,
Acceptability of the protocol and the intervention | At the end of the intervention (+ 12 weeks)
  The acceptability of the protocol and the intervention will be qualitatively assessed through 5 to 7 semi-structured discussion groups by teleconference via the zoom platform. The participants will be interviewed for 75 minutes in sub-groups of 6 to 8 participants on their perception, opinion and experience regarding the intervention and the implementation of the protocol (barriers, facilitators, satisfaction, perceived benefits, recommendation and improvement). An interview guide constructed for the purpose of the study will ensure consistency of the themes explored between the different groups while guiding the group facilitation.

SECONDARY OUTCOMES:
Social physical anxiety change (0-12 weeks) | Before and after intervention (Baseline and after 12 weeks)
  Social physical anxiety scale (validated questionnaire)
Adherence to the physical activity (PA) intervention | At the end of the PA intervention (after 12 weeks)
  Adherence to the PA intervention will be calculated as a percentage from the total number of sessions performed out of the 36 prescribed sessions (frequency).
Compliance with the PA intervention | At the end of the PA intervention (after 12 weeks)
  Compliance with the PA intervention will be calculated as a percentage from the number of sessions for which the participant will have prescribed the prescription compared to all sessions. For these calculations, data from heart rate monitors worn by participants during PA sessions and diaries completed by participants and the kinesiologist will be used.
Physical activity change (0-12 weeks) | Before and after intervention (Baseline and after 12 weeks)
  Triaxial accelerometer (Actigraph® wGT3X-BT) worn on the hip for 7 days
Persistance in the practice of PA after the intervention | Immediately after the intervention and at the end of the study (after 12 weeks and 36 weeks)
  Triaxial accelerometer (Actigraph® wGT3X-BT) worn on the hip for 7 days

OTHER OUTCOMES:
Propensity to immersion | Before the intervention (baseline)
  Validated questionnaire
The feeling of presence in immersion the feeling of presence in immersion | after each virtual reality session (weeks 1, 2, 3, 4, 5,6 , 9 amd 12)
  Gatineau presence questionnaire
Cybermalaise | before and after each virtual reality session (weeks 1, 2, 3, 4, 5,6 , 9 amd 12)
  Simulator Sickness Questionnaire
Sociodemographic data | before the intervention (baseline)
  age, sex,ethnocultural group, level of education, professional status
Depressive symptoms | before the intervention (baseline)
  Center Epidémiologic Scale-Depression-French ; scale (0-3) score range (0-60) higher score = higher depressive symptoms
Food disorder | before the intervention (baseline)
  Eating Attitudes Test-26 ; scale (0-3) score range (0-78), Higher scores indicating greater risk of an eating disorder
Weight Bias Internalisation change (0-12 weeks) | Before and after intervention (Baseline and after 12 weeks)
  Modified Weight Bias Internalisation Scale, scale (1-7), range score (11-77), higher score = higher Weight Bias Internalization)
Body composition change (0-12 weeks) | Before and after intervention (Baseline and after 12 weeks)
  bio-impedance balance (Tanita MC 780U) made by research assistant
Body index mass change (0-12 weeks) | Before and after intervention (Baseline and after 12 weeks)
  scale and measuring rod to measure the size made by research assistant
Waist circumference change (0-12 weeks) | Before and after intervention (Baseline and after 12 weeks)
  tape measure made by research assistant
Body Appreciation change (0-12 weeks) | Before and after intervention (Baseline and after 12 weeks)
  Body Appreciation Scale-2, scale (1-5) score range (1-5), higher score = higher body satisfaction
Perceived pleasure in physical activity in general (0-12 weeks) | Before and after intervention (Baseline and after 12 weeks)
  Physical Activity Enjoyment Scale, scale (1-7) score (1-7) higher score = higher enjoyment
Motivation change (0-12 weeks) | Before and after intervention (Baseline and after 12 weeks)
  Behavioural Regulation In Exercise Questionnaire, scale (0-4), Higher, positive scores indicate greater relative autonomy; lower, negative scores indicate more controlled regulation.
Affects during exercise change (0-12 weeks) | Before and after intervention (Baseline and after 12 weeks)
  Felt Arousal Scale (score 1-6) higher score = higher felt arousal + Feeling Scale (score -5,5) higher score higher pleasure
Self-efficacy change (0-12 weeks) | Before and after intervention (Baseline and after 12 weeks)
  Self efficacy scale (Bandura), scale (0-100) score range (0-100) higher score = higher self efficacy
Perception effort change (0-12 weeks) | Before and after intervention (Baseline and after 12 weeks)
  Borg scale, scale and score range (0-10), higher score = higher perception of effort

CONTACTS AND LOCATIONS:
Locations (1):
- UQO, Gatineau, Quebec, Canada